CLINICAL TRIAL: NCT00643136
Title: Pregabalin BID Add-on Trial: a Randomized, Double-Blind, Placebo-Controlled Parallel-Group Single-Center Sleep EEG Study in Patients With Partial Seizures and Sleep Disturbance Part B: a Randomized, Double-Blind, Placebo-Controlled Parallel-Group Study of Pregabalin Add-on Treatment
Brief Title: A Study of Lyrica as Treatment for Sleep Problems in Patients With Sleep Problems and Seizures
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1008-000-167
Record Dates: First submitted 2008-03-19; First posted 2008-03-26 (Estimated); Last update posted 2008-04-24 (Estimated); Status verified 2008-04

CONDITIONS: Sleep Deprivation; Epilepsies, Partial
MeSH Terms: conditions — Sleep Deprivation; Epilepsies, Partial | interventions — Pregabalin

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Pregabalin (Experimental)
  Interventions: Drug: Pregabalin
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pregabalin — Pregabalin capsules 75 mg twice daily on Days 1-4, then 150 mg twice daily on Days 5-28
  Arms: Pregabalin
Drug: Placebo — Matching placebo capsules twice daily for 28 days
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the effects of pregabalin on sleep problems in patients with seizures.

ELIGIBILITY:
Inclusion Criteria:

* Partial epileptic seizures
* Not taking more than 1 background antiepileptic drug at study entry
* Disturbed sleep

Exclusion Criteria:

* More than 1 secondarily generalized tonic/clonic seizure per week on average over the previous 3 months
* Medical, psychological, or social conditions that could interfere with normal sleep

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2002-11; Study Completion 2004-06 (Actual)

PRIMARY OUTCOMES:
Change from baseline in polysomnographic (PSG) sleep efficiency in the efficacy evaluable population | Endpoint

SECONDARY OUTCOMES:
Change from baseline in total sleep time | Endpoint
Change from baseline in sleep onset latency | Endpoint
Change from baseline in wake after sleep onset | Endpoint
Change from baseline in percent sleep spent in stages 3 and 4 | Endpoint
Change from baseline in percent sleep spent in REM stage | Endpoint
Change from baseline in night sleep quality based on Groningen Sleep Questionnaire (GSQ) | Endpoint
Change from baseline in 4-week sleep quality (Medical Outcomes Study [MOS] Sleep Scale) | Endpoint
Adverse events and laboratory value changes | Endpoint

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (2):
- Netherlands (2):
  - Pfizer Investigational Site, Heeze
  - Pfizer Investigational Site, The Hague

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=1008-000-167&StudyName=A%20study%20of%20Lyrica%20as%20treatment%20for%20sleep%20problems%20in%20patients%20with%20sleep%20problems%20and%20seizures